CLINICAL TRIAL: NCT00847457
Title: Exercise Treatment for Depressed Youth
Brief Title: Depressed Adolescents Treated With Exercise (The DATE Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Carroll Hughes, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH075762 (NIH); R34MH075762 (NIH); DSIR 84-CTCT
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Depression
Keywords: Exercise; Stretching; Adolescents
MeSH Terms: conditions — Depression; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerobic exercise (Experimental): Participants will perform aerobic exercise regularly for 12 weeks.
  Interventions: Behavioral: Aerobic exercise
- Stretch (Active Comparator): Participants will stretch regularly for 12 weeks.
  Interventions: Behavioral: Stretching

INTERVENTIONS:
Behavioral: Aerobic exercise — Aerobic exercises completed three to four times per week for 20 to 30 minutes per session
  Arms: Aerobic exercise
Behavioral: Stretching — Easy to moderate stretching routines completed three times per week, with a new set of routines given each week
  Arms: Stretch

SUMMARY:
This study will evaluate whether standardized aerobic exercise is an effective treatment for depression in adolescents.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a disabling form of depression in which sadness and inability to feel pleasure prevent people from living their normal lives. MDD is common in adolescents, and depression experienced early in life can lead to long-term psychological and social impairment or suicide. Studies of depressed adults show that regular aerobic exercise can result in recovery from mild to moderate MDD. Studies also show that adolescents who exercise regularly have lower rates of depression, but no randomized, controlled studies have examined exercise as a treatment for depression in adolescents. This study will compare a standardized aerobic exercise routine to a stretching control group to determine whether aerobic exercise is an effective treatment for MDD in adolescents.

Participation in this study will last 12 weeks, with follow-up interviews taking place after 6 and 12 months. Participants will first undergo screening procedures, during which adolescent participants and their parents will complete interviews and questionnaires about the adolescent's mood and behavior. Participants will also need to provide physician-written letters confirming that they are healthy enough to participate in the exercise program. After screening, participants will be randomly assigned to either an exercise program or a stretching program. At the first study visit, a course of exercise or stretching will be set for each participant. Participants in both groups will spend the same amount of time doing physical activity. They will complete three to four exercise or stretching sessions per week for 12 weeks, with each session lasting 20 to 30 minutes. Participants will be able to complete some sessions at home, but they will need to return to the study exercise center for weekly study visits. At these study visits, participants will be weighed to determine if the level of exercise needs to be adjusted, and they will complete questionnaires about their depression. Over the course of the study, participants will wear a wrist-watch-like device called an Actical, which will monitor energy use. Participants will also undergo heart rate monitoring while exercising and complete an exercise log online. A set of questionnaires and interviews similar to those at screening will also be repeated at 6- and 12-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of nonpsychotic major depressive disorder at least 4 weeks prior to study entry
* Clinical Global Impression-Severity (CGI-S) score of 4 or greater
* Children's Depression Rating Scale (CDRS) score of greater than 35 but less than 71
* Currently attending school
* Willing and able to use acceptable methods of contraception, if applicable
* A signed letter from family physician verifying physical health necessary for participation in the exercise program
* Response to the Physical Activity Readiness Questionnaire (PAR-Q) indicates that no conditions are present that would render exercise inappropriate
* Speaks and reads English
* Parent or guardian willing to provide informed consent, if applicable

Exclusion Criteria:

* Severe suicidal ideation
* History of psychotic disorders
* Alcohol or substance abuse or dependence within 6 months of study entry
* History of anorexia nervosa or bulimia
* Chronic medical illness requiring regular medication
* Pregnant
* Currently participating in a vigorous exercise program or activity, defined as 30 minutes of vigorous physical activity five times per week
* IQ less than 70

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Childrens Depression Rating Scale - Revised (CDRS-R) | Measured after 12 weeks, 6 months, and 12 months

SECONDARY OUTCOMES:
Exercise feasibility and adherence | Measured after 12 weeks
Amount of energy expended, as measured by the Actical monitor | Measured after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carroll W. Hughes, PhD, ABPP, Principal Investigator — University of Texas Southwestern Medical Center - Dallas

REFERENCES:
- [Background] Hughes CW, Trivedi MH, Cleaver J, Greer TL, Emslie GJ, Kennard B, Dorman S, Bain T, Dubreuil J, Barnes C. DATE: Depressed adolescents treated with exercise: Study rationale and design for a pilot study. Ment Health Phys Act. 2009 Dec;2(2):76-85. doi: 10.1016/j.mhpa.2009.09.005. PMID 20454641